CLINICAL TRIAL: NCT07277114
Title: Drug Coated Balloons Versus Drug-Eluting Stents for Severe Coronary Calcification After Optimal Calcium Modification Assessed by QFR
Brief Title: DCB vs DES for Severe Coronary Calcification After Optimal Modification Assessed by QFR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Tenth People's Hospital affiliated to Tongji University (Unknown)
Responsible Party: Principal Investigator, Junbo Ge, Professor of Medicine/Cardiology and Director of the Department of Cardiology at Zhongshan Hospital, Fudan University,Chairman of the Shanghai Institute of Cardiovascular Diseases., Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025283
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Coronary Calcification
Keywords: coronary calcification; Drug coated balloon; quantitative flow reserve
MeSH Terms: interventions — Atherectomy, Coronary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug coated balloon (Experimental): Drug coated balloon treatment after optimal calcium modification assessed by QFR
  Interventions: Device: rotational atherectomy (RA); Device: excimer laser coronary angioplasty (ELCA); Device: Intravascular Lithotripsy (IVL)
- Drug eluting stent (Active Comparator): Drug eluting stent treatment after optimal calcium modification assessed by QFR
  Interventions: Device: rotational atherectomy (RA); Device: excimer laser coronary angioplasty (ELCA); Device: Intravascular Lithotripsy (IVL)

INTERVENTIONS:
Device: rotational atherectomy (RA) — Rotational atherectomy (RA) is a procedure that uses a diamond-coated, high-speed rotating burr to shave and remove calcified plaque from coronary arteries
Device: excimer laser coronary angioplasty (ELCA) — Excimer laser coronary angioplasty (ELCA) is a minimally invasive procedure that uses pulses of ultraviolet light to vaporize plaque in a blocked coronary artery. The procedure involves inserting a catheter with a laser fiber optic tip into an artery in the groin or arm, guiding it to the blockage using X-ray guidance, and then using the laser to ablate the plaque and improve blood flow.
Device: Intravascular Lithotripsy (IVL) — An IVL catheter with emitters is inserted into the artery, and it delivers pulsatile shock waves to crack the calcium, which then allows for a balloon or stent to be safely expanded to restore blood flow.

SUMMARY:
The goal of this clinical trial is to learn if the short and long term effect of drug coated balloon (DCB) is non-inferior to drug eluting stent (DES) in patients with severe coronary calcification after optimal calcium modification assessed by quantitative flow ratio (QFR). The main questions it aims to answer are:

1. Researchers will compare to see if DCB is non-inferior to DES when evaluated by major cardiovascular adverse events (MACE) one year after percutaneous coronary intervention (PCI).
2. Researchers will compare to see if the perioperative cardiovascular events is different between DCB and DES treated lesions.
3. Researchers will compare to see if the QFR is different between DCB and DES treated lesions one year after PCI.

Participants with severe coronary calcification diagnosed by coronary angiography or intravascular ultrasound (IVUS) will receive calcium modification through rotational atherectomy (RA), excimer laser coronary angioplasty (ELCA), or intravascular lithotripsy (IVL). Then, QFR will be measured based on angiographic image. QFR >0.8 will be defined as optimal calcium modification and patients will be randomized 1:1 to DCB or DES treated groups. Telephone follow-ups will be conducted at 1 month, 6 months after PCI and .angiophraphy follow-up will be performed at 12 months after PCI.

DETAILED DESCRIPTION:
Perioperative cardiovascular events include side branch loss, coronary perforation, no-reflow/slow flow, and perioperative myocardial infarction defined as an elevation of cardiac markers (cTN or CK-MB) greater than 5 times the upper limit of normal.

Definite or probable thrombosis in DCB or DES treated vessels will be documented.

After randomization, if a dissection with restricted blood flow occurs after DCB treatment, DES will be implanted.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

  * Moderate to severe calcified lesions assessed by coronary angiography

    * In situ coronary artery calcification

      * Target lesion with indications for coronary intervention

        * Target lesion vessel diameter ≥ 2.25 mm and ≤ 4.0 mm

          * Calcification modification treatment performed using rotational atherectomy, intravascular lithotripsy (IVL), or excimer laser coronary angioplasty (ELCA).

            * QFR > 0.8 after calcification modification

Exclusion Criteria:

* Patients with ST-segment elevation myocardial infarction:

  * Patients with renal failure requiring dialysis or currently undergoing dialysis.

    * Patients whose coronary angiography quality is unsuitable for QFR analysis.

      * Patients with in-stent restenosis.

        ⑤ Patients with other medical conditions and a life expectancy of <1 year.

        ⑥ Patients scheduled for surgery within 6 months post-procedure, and whose surgery would interfere with continued use of antiplatelet therapy.

        ⑦ Patients who cannot tolerate dual antiplatelet therapy.

        ⑧ Patients who cannot adhere to the protocol-required follow-up, or whose participation in the trial is deemed risky by the investigator.

        ⑨ Patients who cannot provide written informed consent or cannot follow the trial protocol.

        ⑩ Patients currently participating in another clinical trial for coronary interventional devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with MACE as defined by cardiovascular death, target lesion revascularization, non-fatal stroke, target vessel non-fatal myocardial infarction. | One year after treatement.

SECONDARY OUTCOMES:
Perioperative cardiovascular events include side branch loss, coronary perforation, no-reflow/slow flow, and perioperative myocardial infarction defined as an elevation of cardiac markers (cTN or CK-MB) greater than 5 times the upper limit of normal. | From treatment to hospital discharge
QFR at one year post PCI | one year after treatment

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Joh HS, Kwon W, Shin D, Lee SH, Hong YJ, Hong D, Lee SY, Park H, Kim S, Lee SY, Koh JS, Kim H, Kim CJ, Choo EH, Yoon HJ, Park SD, Jeon KH, Bae JW, Ahn SG, Kim SE, Choi KH, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Gwon HC, Lee JM. Drug-Coated Balloon Angioplasty in Patients Undergoing Complex Percutaneous Coronary Intervention. JACC Asia. 2024 Jun 18;4(7):519-531. doi: 10.1016/j.jacasi.2024.04.007. eCollection 2024 Jul. PMID 39101114
- [Result] Muramatsu T, Kozuma K, Tanabe K, Morino Y, Ako J, Nakamura S, Yamaji K, Kohsaka S, Amano T, Kobayashi Y, Ikari Y, Kadota K, Nakamura M; Task Force of the Japanese Association of Cardiovascular Intervention, Therapeutics (CVIT). Clinical expert consensus document on drug-coated balloon for coronary artery disease from the Japanese Association of Cardiovascular Intervention and Therapeutics. Cardiovasc Interv Ther. 2023 Apr;38(2):166-176. doi: 10.1007/s12928-023-00921-2. Epub 2023 Feb 27. PMID 36847902
- [Result] Shin ES, Bang LH, Jun EJ, Her AY, Chung JH, Garg S, Lee JM, Doh JH, Nam CW, Koo BK, Tang Q. Provisional drug-coated balloon treatment guided by physiology on de novo coronary lesion. Cardiol J. 2021;28(4):615-622. doi: 10.5603/CJ.a2020.0105. Epub 2020 Aug 13. PMID 32789835
- [Result] Guedeney P, Claessen BE, Mehran R, Mintz GS, Liu M, Sorrentino S, Giustino G, Farhan S, Leon MB, Serruys PW, Smits PC, von Birgelen C, Ali ZA, Genereux P, Redfors B, Madhavan MV, Ben-Yehuda O, Stone GW. Coronary Calcification and Long-Term Outcomes According to Drug-Eluting Stent Generation. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1417-1428. doi: 10.1016/j.jcin.2020.03.053. PMID 32553329